CLINICAL TRIAL: NCT03549923
Title: Impact of Early CRRT Intervention in Patients Receiving VA-ECMO Support on 30-day Mortality: A Randomized Controlled Trial
Brief Title: Evaluation of Early CRRT InTerventions in Patients With ECMO(ELITE)
Acronym: ELITE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Jianzeng Dong, Director of Heart Failure Center, Beijing Anzhen Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2016YFC1301000
Record Dates: First submitted 2018-05-27; First posted 2018-06-08 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Cardiogenic Shock
Keywords: extracorporeal membrane oxygenation; renal replacement therapy; beta-blocker
MeSH Terms: conditions — Shock, Cardiogenic | interventions — esmolol; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Simultaneous CRRT group (Experimental): CRRT is initiated simultaneously (not late than 24 hours from the initiation of ECMO treatment), regardless of presentation of conventional indication of CRRT. CRRT lasts for 12 hours or more is recommended.The physician can decide when to withdraw CRRT based on the patient's condition.
  Interventions: Device: Simultaneous CRRT
- Conventional-indication CRRT group (Experimental): CRRT is not initiated unless conventional indication of CRRT is presented. The conventional indication of CRRT is as follow: KDIGO stage 3 AKI and one of the following criteria is met: severe hyperkalemia (> 6.5 mmol/L), metabolic acidosis (pH < 7.2), pulmonary edema, blood urea nitrogen level >112 mg/dL, or oliguria (urine output < 200 mL/12 h) for more than 72 hours.
  Interventions: Device: Conventional-indication CRRT
- Esmolol group (Experimental): Patients will receive a continuous esmolol infusion in addition to routine management. The esmolol infusion commences at 25 mg/h and increases by 25 mg/h every 20-minute until the maximal tolerate dosage is reached or the heart rate reduced to 75±5 bpm, or an upper dose limit of 2000 mg/h is reached. Continue infusing esmolol to maintain the heart rate threshold or at the discretion of the physician until either ICU discharge or death. Oral beta-blockers should be considered before the withdrawal of esmolol.
  Interventions: Drug: Esmolol
- Control group (Experimental): All beta-blockers, including esmolol, should not be used during ICU treatment, unless the doctor thinks there's a strong indication.
  Interventions: Drug: Standard care

INTERVENTIONS:
Device: Simultaneous CRRT — The patients in the simultaneous CRRT group will receive CRRT within 24 hours after the initiation of ECMO support.
  Arms: Simultaneous CRRT group
Device: Conventional-indication CRRT — The patients in the conventional-indication group will not receive CRRT until the patient demonstrates AKI and fulfills any one of the criteria of the conventional CRRT indication.
  Arms: Conventional-indication CRRT group
Drug: Esmolol — The patients in esmolol group will receive a continuous esmolol infusion in addition to the standard care.
  Arms: Esmolol group
Drug: Standard care — The patients in control group will not receive any beta-blockers, including esmolol, unless the doctor thinks there's a strong indication.
  Arms: Control group

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is of great value in supporting patients with cardiac shock. More than 80% ECMO patients will develop renal catastrophe that continuous renal replacement therapy (CRRT) is required. The evidence is conflict as to whether early CRRT improves outcomes. Early CRRT before a definite indication developed may prevent side effects of toxicity and fluid overload and therefore, bring survival benefit for the patient. This hypothesis need to be tested in RCT.

Plasma catecholamine levels can be very high in patients under VA-ECMO, which maybe toxic to the cardiac myocardium. Beta-blockers can antagonize the effects of catecholamine. In patients with VA-ECMO, the protective effect of beta-blocker may improve the patients' outcome. This hypothesis also need to be tested in RCT.

ELITE (Evaluation of Early CRRT and Beta-blocker InTerventions in Patients with ECMO) study is a factorial designed RCT with the purpose to test the benefit of early CRRT and beta-blocker in patients treated with V-A ECMO. In the CRRT arm, patients will be randomized to simultaneous CRRT (not late than 24 hours after the initiation of ECMO) or routine therapy (CRRT when indicated). In the beta-blocker arm, patients will be randomized to beta-blocker treatment with a heart rate target of 75±5 bpm or routine therapy. The primary outcome is all-cause mortality at 30 days. Patients discharged alive will be followed for 1 year. Data of mortality and quality of life which are secondary outcomes of this study, will be collected.

DETAILED DESCRIPTION:
Background:

Extracorporeal membrane oxygenation (ECMO) is of great value in supporting patients with severe cardiopulmonary failure, but the mortality rate is still high.

Acute kidney injury (AKI) and fluid overload (FO) are the leading causes of death in patients under Veno-arterial (VA) ECMO. Continuous renal replacement therapy (CRRT) is an effective way to remove toxic substances and provide fluid management. According to current guidelines, CRRT is withhold until at least one of the following criteria is met: severe hyperkalemia (> 6.5 mmol/L), metabolic acidosis (pH < 7.2), pulmonary edema, blood urea nitrogen level > 112 mg/dL, or oliguria (urine output < 200 mL/12h) for more than 72 hours. However, fluid overload and metabolic disorders may cause irreversible damage to the patient and therefore increase mortality. The hypothesis of ELITE study is that simultaneous CRRT may provide better fluid management and avoid metabolic disorders, and bring survival benefit in VA-ECMO patients.

Patients under VA-ECMO are critically ill with high plasma catecholamine levels and treatment of various inotropic agents, which are toxic to the failed myocardium. Beta-blockers can antagonize the effects of endogenous and exogenous catecholamines. The hypothesis of ELITE study is that beta-blocker may protect the failing heart function and reduce 30-day mortality.

Study design:

ELITE study is a prospective, multi-centered, open, 2×2 factorial randomized controlled clinical trial.

In the simultaneous CRRT versus conventional-indication CRRT arm, patients under VA-ECMO will be randomized to the following 2 groups:

1. Simultaneous CRRT group: CRRT is initiated simultaneously (not late than 24 hours from the initiation of ECMO treatment), regardless of presentation of conventional indication of CRRT. CRRT lasts for 12 hours or more is recommended.The physician can decide when to withdraw CRRT based on the patient's condition.
2. Conventional-indication CRRT group: CRRT is not initiated unless conventional indication of CRRT is presented. The conventional indication of CRRT is as follow: KDIGO stage 3 AKI and one of the following criteria is met: severe hyperkalemia (> 6.5 mmol/L), metabolic acidosis (pH < 7.2), pulmonary edema, blood urea nitrogen level >112 mg/dL, or oliguria (urine output < 200 mL/12 h) for more than 72 hours.

In the Beta-blocker versus routine therapy arm, patients with a maintaining dosage of dopamine/dobutamine <5 μg/kg/min, and with neither epinephrine nor norepinephrine will be randomized to the following 2 groups:

1. Esmolol group: Patients will receive a continuous esmolol infusion in addition to routine management. The esmolol infusion commences at 25 mg/h and increases by 25 mg/h every 20-minute until the maximal tolerate dosage is reached or the heart rate reduced to 75±5 bpm, or an upper dose limit of 2000 mg/h is reached. Continue infusing esmolol to maintain the heart rate threshold or at the discretion of the physician until either ICU discharge or death. Oral beta-blockers should be considered before the withdrawal of esmolol.
2. Control group: All beta-blockers, including esmolol, should not be used during ICU treatment, unless the doctor thinks there's a strong indication.

Primary outcome: All-cause mortality at 30 days.

Secondary outcomes:

1. All-cause mortality at 365 days
2. Proportion of patients with long-term RRT indicated
3. Success rate of weaning from ECMO: defined as survive > 24 hours after weaning
4. Any serious adverse events (SAEs), including bleeding, severe arrhythmias, ventilator associated pneumonia, hemorrhagic infection, surgical site infection, any reason induced limb ischemia, stroke and any adverse events that the physician regards as serious.
5. EQ-5D score at 365 days
6. Duration stay at ICU and hospital.
7. Unplanned readmission to hospital.
8. Cause-specific mortality

Sample size consideration:

The sample size calculations are based on the following hypothesis: (a) an estimate 30-day mortality of 70% in the control group; (b) a 20% relative risk reduction for each intervention alone (simultaneous CRRT and beta-blocker); (c) no loss to follow-up; (d) no interaction of the two interventions.

For each intervention, we calculated that a sample size of 496 patients would be required, 248 patients for the treatment group and 248 patients for the control group. In the 2 × 2 factorial design, patients will be randomized to one of four arms, the sample size of each would be 124 patients. With a crossover rate of 10%, the study will randomize 548 patients, 137 patients per arm.

ELIGIBILITY:
Inclusion Criteria for CRRT Study:

1. Patients receiving VA-ECMO support for any reason no longer than 24 hours
2. Provision of informed consent

Exclusion Criteria for CRRT Study:

1. Age < 18 years
2. Patients with convention indication of CRRT: AKI prior to enrollment caused by any reason, at least one of the following criteria is met: severe hyperkalemia (> 6.5 mmol/L), metabolic acidosis (pH < 7.2), pulmonary edema, blood urea nitrogen level > 112 mg/dL, or oliguria (urine output < 200 mL/12h) for more than 72 hours.
3. CKD with estimated GFR<30 mL/min
4. Have already initiated CRRT
5. Active hemorrhage/thrombotic thrombocytopenic purpura
6. Respiratory failure has already initiated VV-ECMO or extracorporeal carbon dioxide removal device before the initiation of VA-ECMO of this time.
7. Prepared for heart transplant or patients received heart transplant.

Inclusion Criteria for Beta-blocker Study:

1. Patients receiving VA-ECMO support for any reason.
2. Dopamine/dobutamine <5 μg/kg/min, no administration of adrenaline or norepinephrine.
3. Within 7 days after initiation of VA-ECMO

Exclusion Criteria for Beta-blocker Study:

1. Age < 18 years
2. Contraindications or intolerance to beta-blockers

   * Moderate or severe bronchial asthma attack or history of bronchial asthma
   * Sinus bradycardia (heart rate < 60 bpm)
   * Type II second-degree or third-degree AVB
   * Allergy to esmolol
3. For women at child bearing age, pregnant or positive pregnancy test.
4. Respiratory failure has already initiated VV-ECMO or extracorporeal carbon dioxide removal device before the initiation of VA-ECMO of this time
5. Have been on beta-blocker treatment after initiation of ECMO
6. Prepared for heart transplant or patients received heart transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 days

SECONDARY OUTCOMES:
All-cause mortality | 365 days
Proportion of patients receiving long-term RRT | 365 days/when patient dies
Success rate of weaning from ECMO | 30 days
  Success weaning from ECMO is defined as survive > 24 hours after weaning
Any serious adverse events (SAEs) | 30 days
  Including bleeding, severe arrhythmias, ventilator associated pneumonia, hemorrhagic infection, surgical site infection, any reason induced limb ischemia, stroke and any adverse events that the physician regards as serious.
EQ-5D score | 365 days
Duration stay at ICU and hospital | 365 days
Unplanned readmission to hospital | 30 days
Cause-specific mortality | 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Jianzeng Dong, PhD., Md., Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Werdan K, Muller U, Reithmann C, Pfeifer A, Hallstrom S, Koidl B, Schlag G. Mechanisms in acute septic cardiomyopathy: evidence from isolated myocytes. Basic Res Cardiol. 1991 Sep-Oct;86(5):411-21. doi: 10.1007/BF02190709. PMID 1662946
- [Background] Aso S, Matsui H, Fushimi K, Yasunaga H. In-hospital mortality and successful weaning from venoarterial extracorporeal membrane oxygenation: analysis of 5,263 patients using a national inpatient database in Japan. Crit Care. 2016 Apr 5;20:80. doi: 10.1186/s13054-016-1261-1. PMID 27044572
- [Background] Chen H, Yu RG, Yin NN, Zhou JX. Combination of extracorporeal membrane oxygenation and continuous renal replacement therapy in critically ill patients: a systematic review. Crit Care. 2014 Dec 8;18(6):675. doi: 10.1186/s13054-014-0675-x. PMID 25482187
- [Background] Alonso de Vega JM, Diaz J, Serrano E, Carbonell LF. Oxidative stress in critically ill patients with systemic inflammatory response syndrome. Crit Care Med. 2002 Aug;30(8):1782-6. doi: 10.1097/00003246-200208000-00018. PMID 12163793
- [Background] Bohm M, Link A, Cai D, Nieminen MS, Filippatos GS, Salem R, Cohen Solal A, Huang B, Padley RJ, Kivikko M, Mebazaa A. Beneficial association of beta-blocker therapy on recovery from severe acute heart failure treatment: data from the Survival of Patients With Acute Heart Failure in Need of Intravenous Inotropic Support trial. Crit Care Med. 2011 May;39(5):940-4. doi: 10.1097/CCM.0b013e31820a91ed. PMID 21283007
- [Background] Rudiger A. Beta-block the septic heart. Crit Care Med. 2010 Oct;38(10 Suppl):S608-12. doi: 10.1097/CCM.0b013e3181f204ca. PMID 21164404
- [Background] Sander O, Welters ID, Foex P, Sear JW. Impact of prolonged elevated heart rate on incidence of major cardiac events in critically ill patients with a high risk of cardiac complications. Crit Care Med. 2005 Jan;33(1):81-8; discussion 241-2. doi: 10.1097/01.ccm.0000150028.64264.14. PMID 15644652
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Champion S, Belcour D, Vandroux D, Drouet D, Gauzere BA, Bouchet B, Bossard G, Djouhri S, Jabot J, Champion M, Lefort Y. Stress (Tako-tsubo) cardiomyopathy in critically-ill patients. Eur Heart J Acute Cardiovasc Care. 2015 Apr;4(2):189-96. doi: 10.1177/2048872614547686. Epub 2014 Sep 8. PMID 25202025
- [Background] Yan X, Jia S, Meng X, Dong P, Jia M, Wan J, Hou X. Acute kidney injury in adult postcardiotomy patients with extracorporeal membrane oxygenation: evaluation of the RIFLE classification and the Acute Kidney Injury Network criteria. Eur J Cardiothorac Surg. 2010 Feb;37(2):334-8. doi: 10.1016/j.ejcts.2009.07.004. Epub 2009 Aug 18. PMID 19692267
- [Background] Isogai T, Matsui H, Tanaka H, Fushimi K, Yasunaga H. Early beta-blocker use and in-hospital mortality in patients with Takotsubo cardiomyopathy. Heart. 2016 Jul 1;102(13):1029-35. doi: 10.1136/heartjnl-2015-308712. Epub 2016 Feb 15. PMID 26879240
- [Background] Andreis DT, Singer M. Catecholamines for inflammatory shock: a Jekyll-and-Hyde conundrum. Intensive Care Med. 2016 Sep;42(9):1387-97. doi: 10.1007/s00134-016-4249-z. Epub 2016 Feb 12. PMID 26873833
- [Background] Salvadori A, Pasquier P, Jarrassier A, Renner J, Merat S. Adverse cardiac events during catecholamine therapy: a role for hydrocortisone? Intensive Care Med. 2012 Oct;38(10):1725; author reply 1726. doi: 10.1007/s00134-012-2663-4. Epub 2012 Aug 7. No abstract available. PMID 22868276
- [Background] Schmidt M, Bailey M, Kelly J, Hodgson C, Cooper DJ, Scheinkestel C, Pellegrino V, Bellomo R, Pilcher D. Impact of fluid balance on outcome of adult patients treated with extracorporeal membrane oxygenation. Intensive Care Med. 2014 Sep;40(9):1256-66. doi: 10.1007/s00134-014-3360-2. Epub 2014 Jun 17. PMID 24934814
- [Background] Schmittinger CA, Torgersen C, Luckner G, Schroder DC, Lorenz I, Dunser MW. Adverse cardiac events during catecholamine vasopressor therapy: a prospective observational study. Intensive Care Med. 2012 Jun;38(6):950-8. doi: 10.1007/s00134-012-2531-2. Epub 2012 Apr 12. PMID 22527060
- [Background] Chen YC, Tsai FC, Fang JT, Yang CW. Acute kidney injury in adults receiving extracorporeal membrane oxygenation. J Formos Med Assoc. 2014 Nov;113(11):778-85. doi: 10.1016/j.jfma.2014.04.006. Epub 2014 Jun 10. PMID 24928419
- [Background] Dunser MW, Hasibeder WR. Sympathetic overstimulation during critical illness: adverse effects of adrenergic stress. J Intensive Care Med. 2009 Sep-Oct;24(5):293-316. doi: 10.1177/0885066609340519. Epub 2009 Aug 23. PMID 19703817
- [Background] Prins KW, Neill JM, Tyler JO, Eckman PM, Duval S. Effects of Beta-Blocker Withdrawal in Acute Decompensated Heart Failure: A Systematic Review and Meta-Analysis. JACC Heart Fail. 2015 Aug;3(8):647-53. doi: 10.1016/j.jchf.2015.03.008. PMID 26251094
- [Background] Morelli A, Ertmer C, Westphal M, Rehberg S, Kampmeier T, Ligges S, Orecchioni A, D'Egidio A, D'Ippoliti F, Raffone C, Venditti M, Guarracino F, Girardis M, Tritapepe L, Pietropaoli P, Mebazaa A, Singer M. Effect of heart rate control with esmolol on hemodynamic and clinical outcomes in patients with septic shock: a randomized clinical trial. JAMA. 2013 Oct 23;310(16):1683-91. doi: 10.1001/jama.2013.278477. PMID 24108526
- [Background] Zarbock A, Kellum JA, Schmidt C, Van Aken H, Wempe C, Pavenstadt H, Boanta A, Gerss J, Meersch M. Effect of Early vs Delayed Initiation of Renal Replacement Therapy on Mortality in Critically Ill Patients With Acute Kidney Injury: The ELAIN Randomized Clinical Trial. JAMA. 2016 May 24-31;315(20):2190-9. doi: 10.1001/jama.2016.5828. PMID 27209269
- [Background] Goldstein SL, Somers MJ, Baum MA, Symons JM, Brophy PD, Blowey D, Bunchman TE, Baker C, Mottes T, McAfee N, Barnett J, Morrison G, Rogers K, Fortenberry JD. Pediatric patients with multi-organ dysfunction syndrome receiving continuous renal replacement therapy. Kidney Int. 2005 Feb;67(2):653-8. doi: 10.1111/j.1523-1755.2005.67121.x. PMID 15673313
- [Background] Annane D, Bellissant E, Cavaillon JM. Septic shock. Lancet. 2005 Jan 1-7;365(9453):63-78. doi: 10.1016/S0140-6736(04)17667-8. PMID 15639681
- [Background] Singer M. Catecholamine treatment for shock--equally good or bad? Lancet. 2007 Aug 25;370(9588):636-7. doi: 10.1016/S0140-6736(07)61317-8. No abstract available. PMID 17719998
- [Background] Gaudry S, Hajage D, Schortgen F, Martin-Lefevre L, Pons B, Boulet E, Boyer A, Chevrel G, Lerolle N, Carpentier D, de Prost N, Lautrette A, Bretagnol A, Mayaux J, Nseir S, Megarbane B, Thirion M, Forel JM, Maizel J, Yonis H, Markowicz P, Thiery G, Tubach F, Ricard JD, Dreyfuss D; AKIKI Study Group. Initiation Strategies for Renal-Replacement Therapy in the Intensive Care Unit. N Engl J Med. 2016 Jul 14;375(2):122-33. doi: 10.1056/NEJMoa1603017. Epub 2016 May 15. PMID 27181456
- [Background] Yap HJ, Chen YC, Fang JT, Huang CC. Combination of continuous renal replacement therapies (CRRT) and extracorporeal membrane oxygenation (ECMO) for advanced cardiac patients. Ren Fail. 2003 Mar;25(2):183-93. doi: 10.1081/jdi-120018719. PMID 12739825
- [Derived] Wang X, Wang H, Du X, Wang Z, Li C, Anderson CS, Zhang J, Hou X, Dong J. EvaLuation of early CRRT and beta-blocker InTervention in patients with ECMO (ELITE) trial: study protocol for a 2 x 2 partial factorial randomized controlled trial. Trials. 2022 Aug 19;23(1):684. doi: 10.1186/s13063-022-06617-x. PMID 35986410